CLINICAL TRIAL: NCT04062669
Title: Safety and Immunogenicity of GSK's Rabies G SAM (CNE) Vaccine [GSK3903133A] in Healthy Adults.
Brief Title: A Study to Evaluate the Safety and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Experimental Rabies Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 208608
Record Dates: First submitted 2019-08-06; First posted 2019-08-20 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Virus Diseases
Keywords: First Time in Human; Vaccine; Healthy subjects; Rabies
MeSH Terms: conditions — Virus Diseases; Rabies | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In Part 1 of the study, only data during the primary vaccination phase (from study start to Day 91) will be collected in an observer-blind manner. By observer-blind, it is meant that the vaccines recipient and those responsible for the evaluation of any study endpoint will all be unaware of which vaccine was administered.
  For Part 1, the study will be observer-blind until Day 91. When the Day 91 analysis will result in unblinding of all the subjects to the sponsor. Therefore, the study cannot be considered observer-blind beyond Day 91 and will be conducted in a single-blind* manner thereafter; with all subjects remaining blinded up to study conclusion (Month 14).
  For Part 2, the study will be conducted in open-label manner from study start to study conclusion.
  *Due to the recent COVID-19 pandemic, the study will be fully unblinded from study start to study conclusion to allow all subject treatments to be known to the team and investigators, thereby facilitating rapid safety assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Low dose (Ld-) RG SAM (CNE) group (Experimental): In Part 1 of the study, healthy adults, 18 to 40 years of age, will receive one intramuscular injection of RG SAM (CNE) low dose formulation vaccine in one arm and one intramuscular injection of saline solution in the opposite arm at Days 1 and 61).
  In Part 2 of the study, healthy adults, 18 to 40 years of age, will receive one intramuscular injection of RG SAM (CNE) low dose formulation vaccine in one arm according to a 0, 2, 6-month schedule (i.e. at Days 1 and 61)
  Interventions: Biological: Low dose formulation of RG SAM (CNE) vaccine (GSK3903133A)
- Medium dose (Md-) RG SAM (CNE) group (Experimental): Healthy adults,18 to 40 years of age, will receive one intramuscular injection of RG SAM (CNE) medium dose formulation vaccine in one arm and one intramuscular injection of saline solution in the opposite arm at Day 1.
  Interventions: Biological: Medium dose formulation of RG SAM (CNE) vaccine (GSK3903133A)
- Lower dose (Lrd-) RG SAM (CNE) group (Experimental): Healthy adults, 18 to 40 years of age, will receive one intramuscular injection of RG SAM (CNE) lower dose formulation vaccine in one arm according to a 0, 2, 6-month schedule (i.e. at Days 1 and 61)
  Interventions: Biological: Lower dose formulation of RG SAM (CNE) vaccine (GSK3903133A)
- Lowest dose (Ltd-) RG SAM (CNE) group (Experimental): Healthy adults, 18 to 40 years of age, will receive one intramuscular injection of RG SAM (CNE) lowest dose formulation vaccine in one arm according to a 0, 2, 6-month schedule (i.e. at Days 1 and 61)
  Interventions: Biological: Lowest dose formulation of RG SAM (CNE) vaccine (GSK3903133A)
- Saline Placebo group (Placebo Comparator): In Part 1 of the study, healthy adults, 18 to 40 years of age, will receive two intramuscular injections of saline placebo, one in each arm, according to a 0, 2, 6-month schedule (i.e. at Days 1 and 61).
  In Part 2 of the study, healthy adults, 18 to 40 years of age will receive one intramuscular injections of saline placebo in one arm according to a 0, 2, 6-month schedule (i.e. at Days 1 and 61).
  Interventions: Drug: Saline Placebo
- RabAvert group (Active Comparator): In Part 1 of the study, healthy adults, 18 to 40 years of age, will receive one intramuscular injection of RabAvert in one arm and one intramuscular injection of saline solution in the other arm, according to a 0, 2, 6-month schedule (i.e. at Days 1 and 61).
  In Part 2 of the study, healthy adults, 18 to 40 years of age, will receive one intramuscular injection of RabAvert in one arm according to a 0, 2, 6-month schedule (i.e. at Days 1 and 61).
  Interventions: Biological: RabAvert

INTERVENTIONS:
Biological: Low dose formulation of RG SAM (CNE) vaccine (GSK3903133A) — Subjects in the low dose (Ld-) RG SAM (CNE) group will receive 2 doses of RG SAM (CNE) low dose formulation, administered intramuscularlyat Days 1 and 61.
  Arms: Low dose (Ld-) RG SAM (CNE) group
Biological: Medium dose formulation of RG SAM (CNE) vaccine (GSK3903133A) — Subjects in the medium dose (Md-) RG SAM (CNE) group will receive 1 doses of RG SAM (CNE) medium dose formulation, administered intramuscularly at Day 1.
  Arms: Medium dose (Md-) RG SAM (CNE) group
Biological: Lower dose formulation of RG SAM (CNE) vaccine (GSK3903133A) — Subjects in the Lower dose (Lrd-) RG SAM (CNE) group will receive 2 doses of RG SAM (CNE) lower dose formulation, administered intramuscularly, according to a 0, 2-month schedule (i.e. at Days 1 and 61)
  Arms: Lower dose (Lrd-) RG SAM (CNE) group
Biological: Lowest dose formulation of RG SAM (CNE) vaccine (GSK3903133A) — Subjects in the Lowest dose (Ltd-) RG SAM (CNE) group will receive 2 doses of RG SAM (CNE) lowest dose formulation, administered intramuscularly, according to a 0, 2-month schedule (i.e. at Days 1 and 61)
  Arms: Lowest dose (Ltd-) RG SAM (CNE) group
Drug: Saline Placebo — Subjects in the Saline Placebo group will receive 2 doses of saline Placebo, administered intramuscularly Day 1 and 61.
  Arms: Saline Placebo group
Biological: RabAvert — Subjects in the RabAvert Group will receive 2 doses of RabAvert vaccine, administered intramuscularly, at Days 1 and 61.
  Arms: RabAvert group

SUMMARY:
The purpose of this first time-in-human (FTiH) study is to evaluate the safety, reactogenicity and immunogenicity of different dose levels of an experimental rabies glycoprotein G (RG) vaccine (RG-SAM [CNE] vaccine), made using a new technology, when administered intramuscularly (IM) on a 0, 2, 6 *-month schedule to healthy adults.

* There will be no vaccinations with the third dose of any of the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. participation in genetics research, completion of the electronic diary cards, return for follow-up visits).
* Written informed consent obtained from the participant prior to performance of any study specific procedure.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* A male or female participant between, and including, 18 and 40 years of age at the time of the first vaccination.
* Body Mass Index >18 Kg/m^2 and <35 Kg/m^2.
* Participants with following hematological/biochemical parameters:

  * White Blood Cells and differential, within the study designated laboratory normal range. Participants with FDA toxicity grade 1 differential cell counts and considered not clinically significant may be enrolled at the discretion of the investigator, and with the review and approval of the medical monitor.
  * Platelets = 125,000 - 500,000 cells/mm^3
  * Hemoglobin within normal range of the study designated laboratory
  * Alanine aminotransferase within the study designated laboratory normal range
  * Aspartate aminotransferase within the study designated laboratory normal range
  * Total bilirubin within the study designated laboratory normal range
  * Alkaline phosphatase within the study designated laboratory normal range
  * Serum creatinine less than or equal to 1.1 times study designated laboratory's upper normal limit .
  * Seronegative for hepatitis B surface antigen, hepatitis C virus antibodies, or human immunodeficiency virus antibodies
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female participants of childbearing potential may be enrolled in the study, if the participant

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series

Exclusion Criteria:

* History of diagnosis with rabies exposure, infection or disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of or current autoimmune disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any components of RabAvert including polygeline, bovine gelatin, neomycin, chlortetracycline and amphotericin B, chicken protein, egg products or any other vaccine component.
* Lymphoproliferative disorder or malignancy within previous 5 years (excluding effectively treated non-melanotic skin cancer).
* Hypersensitivity to latex.
* History of Type I hypersensitivity reactions to any beta-lactam antibiotics (penicillin, aminopenicillins, cephalosporins and carbapenems).
* Any acute or chronic, clinically significant disease, as determined by physical examination, laboratory screening tests, subject personal report and/or General Physician (GP) information.
* Use of any investigational or non-registered product other than the study vaccines during the period starting 30 days before the first dose of study vaccines, or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the vaccination and ending 30 days after (Influenza vaccine excluded).
* Previous vaccination with any licensed or investigational rabies vaccine.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period within 6 months prior to the vaccine dose.
* Current allergy treatment with allergen immunotherapy with antigen injections, unless on maintenance schedule.
* Concomitant or planned administration of antimalarial drugs, to include hydroxychloroquine within 30 days of vaccination.
* Current anti-tuberculosis prophylaxis or therapy.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been/will be exposed to an investigational or a non-investigational vaccine/product.
* Pregnant or lactating female participant.
* Female participant planning to become pregnant or planning to discontinue contraceptive precautions.
* Participants at a higher risk than the average US resident with regard to exposure to rabies, per the RabAvert package insert and rabies vaccination recommendations from the Centers for Disease Control (CDC).
* Participants with extensive tattoos covering deltoid region on both the arms that would preclude the assessment of local reactogenicity.
* Planned move to a location that will prohibit participating in the trial until study end.
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited local adverse events (AEs) during the 7-day follow-up period after the first dose received in the Primary vaccination phase | During the 7-day follow-up period after the first dose (administered at Day 1)
  The following local AEs are solicited: pain, redness and swelling at injection site.
Number of participants reporting solicited local adverse events (AEs) during the 7-day follow-up period after the second dose received in the Primary vaccination phase | During the 7-day follow-up period after the second dose (administered at Day 61)
  The following local AEs are solicited: pain, redness and swelling at injection site.
Number of participants reporting solicited general AEs during the 7-day follow-up period after the first dose received in the Primary vaccination phase | During the 7-day follow-up period after the first dose (administered at Day 1)
  The following general AEs are solicited: fatigue, fever, nausea, vomiting, diarrhea, abdominal pain and headache.
  Fever is defined as temperature ≥ 38.0°C / 100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
Number of participants reporting solicited general AEs during the 7-day follow-up period after the second dose received in the Primary vaccination phase | During the 7-day follow-up period after the second dose (administered at Day 61)
  The following general AEs are solicited: fatigue, fever, nausea, vomiting, diarrhea, abdominal pain and headache.
  Fever is defined as temperature ≥ 38.0°C / 100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
Number of participants reporting unsolicited AEs during a 30-day follow-up period follow-up after the first dose received in the Primary vaccination phase | During the 30-day follow-up period after the first dose (administered at Day 1).
  Unsolicited AE is defined as an AE reported in addition to those solicited during the clinical study and as any solicited AE with onset outside the specified period of follow-up for solicited symptoms.
Number of participants reporting unsolicited AEs during a 30-day follow-up period follow-up after the second dose received in the Primary vaccination phase | During the 30-day follow-up period after the second dose (administered at Day 61).
  Unsolicited AE is defined as an AE reported in addition to those solicited during the clinical study and as any solicited AE with onset outside the specified period of follow-up for solicited symptoms.
Number of participants with hematological and biochemical laboratory abnormalities at Day 1. | At Day 1
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry and hematology) are reported. The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of participants with hematological and biochemical laboratory abnormalities at Day 4. | At Day 4.
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry and hematology) are reported. The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of participants with hematological and biochemical laboratory abnormalities at Day 8. | At Day 8.
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry and hematology) are reported. The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of participants with hematological and biochemical laboratory abnormalities at Day 61. | At Day 61.
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry and hematology) are reported. The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of participants with hematological and biochemical laboratory abnormalities at Day 64. | At Day 64.
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry and hematology) are reported. The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of participants with hematological and biochemical laboratory abnormalities at Day 68. | At Day 68.
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry and hematology) are reported. The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of participants reporting medically attended AE (MAEs) | During 90 days (from Day 1 to Day 91)
  A medically attended adverse event is an AE for which the participants received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (i.e., nurse practitioner or physician assistant or medical doctor) for any reason.
Number of participants reporting serious adverse events (SAEs) | During 90 days (from Day 1 to Day 91)
  SAEs assessed include any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study patient.
Number of participants reporting potential immune-mediated diseases (pIMDs) | During 90 days (from Day 1 to Day 91)
  pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.

SECONDARY OUTCOMES:
Number of participants reporting solicited local adverse events (AEs) during the 7-day follow-up period after each vaccination received from Day 1 up to study conclusion at Month 18 | During the 7-day follow-up period after the third dose (administered at Day 181)
  The following local AEs are solicited: pain, redness and swelling at injection site.
Number of participants reporting solicited general AEs during the 7-day follow-up period after each vaccination received from Day 1 up to study conclusion at Month 18 | During the 7-day follow-up period after the third dose (administered at Day 181)
  The following general AEs are solicited: fatigue, fever, nausea, vomiting, diarrhea, abdominal pain and headache.
  Fever is defined as temperature ≥ 38.0°C / 100.4°F. The preferred location for measuring temperature in this study is the oral cavity.
Number of participants reporting unsolicited AEs during a 30-day follow-up period after each vaccination from Day 1 up to study conclusion at Month 18 | During the 30-day follow-up period after the third dose (administered at Day 181)
  Unsolicited AE is defined as an AE reported in addition to those solicited during the clinical study and as any solicited AE with onset outside the specified period of follow-up for solicited symptoms.
Number of participants with hematological and biochemical laboratory abnormalities at Day 1, Day 4, Day 8, Day 61, Day 64, Day 68, Day 181, Day 184 and Day 188 | At Day 1, Day 4, Day 8, Day 61, Day 64, Day 68, Day 181, Day 184 and Day 188
  Clinically significant abnormal laboratory findings (e.g. clinical chemistry and hematology) are reported. The investigator exercises his or her medical and scientific judgement in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant.
Number of participants reporting MAEs from Day 1 up to study conclusion at Month 14 | From Day 1 up to study conclusion at Month 14
  A medically attended adverse event is an AE for which the participants received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (i.e., nurse practitioner or physician assistant or medical doctor) for any reason.
Number of participants reporting SAEs from Day 1 up to study conclusion at Month 14 | From Day 1 to up to study end at Month 14
  SAEs assessed include any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study patient.
Number of participants reporting pIMDs from Day 1 up to study conclusion at Month 14 | From Day 1 up to study conclusion at Month 14
  pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Evaluation of immunogenicity in terms of Rabies Virus Neutralizing Antibody (RVNA) concentrations | At Day 1 and Day 91
  RVNA concentrations determined by Rapid Fluorescence Foci Inhibition Test (RFFIT) are presented as geometric mean concentrations (GMCs), expressed in International Unit per milliliter (IU/mL).
Evaluation of immunogenicity in terms of Anti-rabies G IgG antibody concentrations | At Day 1 and Day 91
  Anti-rabies G IgG antibody concentrations determined by Enzyme Linked Immunosorbent Assay (ELISA) are presented as GMCs, expressed in ELISA unit per milliliter (EU/mL).
Evaluation of persistence of immunogenicity in terms of anti-rabies G IgG antibody concentrations at 5 months after last vaccination | At Month 7 (i.e. 5 months after the last vaccination)
  Anti-rabies G IgG antibody concentrations determined by ELISA are presented as GMCs, expressed in EU/mL.
Evaluation of persistence of immunogenicity in terms of anti-rabies G IgG antibody concentrations at 10 months after last vaccination | At Month 12 (i.e. 10 months after the last vaccination)
  Anti-rabies G IgG antibody concentrations determined by ELISA are presented as GMCs, expressed in EU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (4):
- United States (4):
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an exemption can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com